CLINICAL TRIAL: NCT05094687
Title: Cutaneous Manifestations of Coronavirus Disease 2019(COVID-19).
Status: Completed | Type: Observational
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Rabia Ghafoor, Rabia ghafoor, Jinnah Postgraduate Medical Centre
Other Study IDs: NO.F.2-81/2021-GEN/61595/JPMC
Record Dates: First submitted 2021-10-23; First posted 2021-10-26 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cutaneous Manifestations; Skin Manifestations; COVID-19; COVID-19 Pneumonia; COVID-19 Pandemic; Corona Virus Infection; Coronavirus Disease 2019; Sars-CoV-2 Infection
Keywords: COVID-19; COVID-19 pneumonia; COVID-19 pandemic; Coronavirus disease 2019; Skin manifestations; Cutaneous manifestations; Cutaneous patterns; Livedo reticularis; Pseudo chilblains; Pernio-like lesion; Chilblains; Maculopapular rash; Scabies; Pityriasis rosea; Acral ischemia; Blue toe; Pustular; Papulopustular; Purpura fulminans; Urticaria; Erythema multiforme; Pruritis; Xerosis; Herpes zoster; Tinea; Papulosquamous; Vasculitis; Pityriasis versicolor; Aphthous ulcer; Oral candidiasis; Vesicular rash
MeSH Terms: conditions — Skin Manifestations; COVID-19; Coronavirus Infections; Livedo Reticularis; Chilblains; Scabies; Pityriasis Rosea; Purpura Fulminans; Urticaria; Erythema Multiforme; Pruritus; Herpes Zoster; Tinea; Vasculitis; Tinea Versicolor; Stomatitis, Aphthous; Candidiasis, Oral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An outbreak of Corona virus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-coV-2) occurred in Wuhan city, Hubei province, China in December 2019. Pulmonary health has been the main focus of studies of COVID-19, current articles show that cutaneous signs appear in COVID-19 patients, their identification may be vital to early diagnosis and lead to possible better prognosis in COVID-19 patients

DETAILED DESCRIPTION:
INTRODUCTION: An outbreak of Corona virus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-coV-2) occurred in Wuhan city, Hubei province, China in December 2019. Although pulmonary health has been the main focus of studies, recent studies show that cutaneous symptoms appear in COVID-19 patients, with differing levels of severity even in those patients who were once thought to be asymptomatic to the infection. Recent studies show association of skin manifestations of COVID-19 with severity of COVID-19 infection, which These days, ongoing interest of clinical trials. Although not much is known concerning the pathophysiologic mechanisms of these cutaneous manifestations, their identification may be vital to early diagnosis and lead to possible better prognosis in COVID-19 patients.

OBJECTIVE: To examine cutaneous manifestations of Coronavirus Disease-19 (COVID-19).

PLACE OF STUDY: Department of Dermatology Jinnah Postgraduate Medical Centre (JPMC) Karachi, Sindh, Pakistan.

RESEARCH METHODOLOGY: The longitudinal study will be conducted on patients with COVID-19 at JPMC Karachi. Permission from the ethical review committee will be taken prior to conduction of study and demographic data and informed consent will be taken from every patient or their guardians. forr data collection non-probability convenience sampling method will be used. Sample size of study would be 1206 polymerase chain reaction (PCR) for SARS-CoV-2 RNA positive patients. Detailed history and examination of patients including cutaneous examination be conducted in COVID-19 patients by dermatologists. The data would include gender, age at the time of onset of COVID-19, presence/ absence of comorbidities, the presence/absence of cutaneous manifestation, cutaneous patterns, the duration of skin manifestations, presence or absence of systemic symptoms, skin-related symptoms, type of systemic symptoms, the duration of systemic symptoms, the time of onset of skin manifestation, the latency between the systemic symptoms and cutaneous manifestations, and the COVID-19 severity ( mild/asymptomatic (gastrointestinal symptoms, cough or fever) moderate (dyspnea or pneumonia on x-ray) or severe (death, thromboembolic event or ventilator). The lab-confirmed COVID-19 patients 20 years of age or older irrespect of symptoms were included. Patients with pre-existing dermatological disease, autoimmune disease, malignancy or chemotherapy, pregnant or lactating women, blood transfusion, on immunosuppressant, malabsorption syndrome or taking any drug/vaccine within 14 days before onset of skin lesions will be excluded. Photographs of skin lesions will be taken by consent.

DATA ANALYSIS: SPSS version 23 registered for Microsoft windows will be used for analysis. Mean and standard deviation will be calculated for expression of quantitative variables like age and disease duration of skin. Systemic symptoms duration, the latency between the systemic and cutaneous manifestations, and age for disease outcome will be calculated by median and interquartile range. Gender, co-morbidities, presence or absence of cutaneous/ systemic manifestations, cutaneous symptoms, skin patterns, time of onset of rash, and disease outcome covid-19 will be calculated by frequencies and percentages. Effect modifiers like age, gender, weight, co-morbidities, duration of symptoms will be controlled through stratification. Poststratification will be recalculated and chi-square test will be applied. P-value of <0.05% will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

both genders Any age PCR diagnosed COVID-19 patient irrespective of symptoms

Exclusion Criteria:

patient with diagnosed case of autoimmune disease on drugs known case of malignancy or chemotherapy recurrent transfusion history diagnosed case of malabsorption syndrome On immunosuppressant. Already having any prior skin disease Any drug/vaccine taken within 14 days before onset of rash Pregnant or lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1206 patients diagnosed case of COVID-19 by PCR.
Sampling Method: Non-Probability Sample
Enrollment: 1206 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Frequency of skin manifestations in 1206 | From day of randomisation until development of skin manifestations or not, assessed upto 12 months
  Frequency of skin manifestations in COVID-19 positive 1206 subjects.
COVID-19 Disease Outcome in patients with skin manifestations | Disease outcome during this 12 months duration of study.
  Disease outcome of COVID-19 in participants who will be having cutanous manifestations and will be classified as mild moderate and severe.
Cutaneous patterns | From day of randomisation until development of skin manifestations or not, assessed upto 12 months
  If present, type of skin manifestations to be noted
Association of COVID-19 disease outcome in correlation with skin manifestation | From day of randomisation until development of skin manifestations or not, until COVID-19 disease outcome (improved, worsen or death) assessed upto 12 months
  It is to check if presence of skin manifestations can affect COVID-19 disease outcome
Skin symptoms | From day of randomisation until development of skin manifestations or not, assessed upto 12 months
  If applicable, Skin symptoms as pruritis, burning or pain
Duration of skin manifestations | From day of randomisation until development of skin manifestation or not, if development/already developed skin manifestations then resolution of it or for how long it persisted, assessed upto 12 months
  For how long the skin manifestations last before resolution or whether it persisted.
The time of onset of skin manifestations | From day of randomisation until development of systemic manifestations or not, in patients with skin manifestations assessed upto 12 months
  To check if skin manifestations can be an early sign of disease or a sole manifestation of COVID-19. (without, before, after or with systemic symptoms)
Presence or absence of systemic symptoms in COVID-19 patients | Day 1 of randomisation until development of systemic symptoms in patients with skin manifestations in upto 12 months
  To check if skin manifestations can be a sole presentation of COVID-19

SECONDARY OUTCOMES:
Latency between the cutaneous manifestations and development of systemic symptoms of COVID-19 | From day of randomisation until development of skin/systemic manifestations or not, assessed upto 12 months
  To check if skin manifestations could be earlier symptom of COVID-19.
Duration of systemic symptoms | From day of randomisation to recovery or death, and also duration of symptoms prior to coming for consultation/hospital, assessed upto 12 months
  Duration of systemic symptoms till recovery or death
Type of systemic symptoms | From day of randomisation until development of systemic symptoms or not, assessed upto 12 months
  To help categorising disease outcomes
age of patients | Day 1 of randomisation until development of skin manifestations in upto 12 months
  to check which category of manifestation occurs more commonly at what age
comorbidities | Day 1 of randomisation until development of skin manifestations in upto 12 months
  to check their affect on disease outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, MBBS, FCPS, SCE-Derm(MRCP-UK), Principal Investigator — Jinnah Postgraduate Medical Centre; Syeda Mahanum Ali, MBBS, Postgraduate Trainee, Principal Investigator — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan